CLINICAL TRIAL: NCT02758977
Title: Associating Liver Partition With Portal Vein Ligation for Staged Hepatectomy (ALPPS) vs. Conventional Two-Stage Hepatectomy (TSH) for Surgical Treatment of Marginally Resectable Colorectal Liver Metastases (CRLM) - A Multicentric, Randomized Controlled Trial
Brief Title: Associating Liver Partition With Portal Vein Ligation for Staged Hepatectomy (ALPPS) vs. Two-Stage Hepatectomy (TSH) for Marginally Resectable Colorectal Liver Metastases (CRLM)
Acronym: ALPPSforCRLM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-0024
Record Dates: First submitted 2016-04-05; First posted 2016-05-03 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Colon Cancer Liver Metastases; Liver Neoplasms; Liver Diseases; Secondary Malignant Neoplasm of Liver; Malignant Neoplasm of Large Intestine Metastatic to Liver; Hepatectomy; Surgery
Keywords: Colorectal liver metastases; Liver Surgery; ALPPS; Two Stage Hepatectomy; Surgical Oncology; Hepatectomy
MeSH Terms: conditions — Liver Neoplasms; Liver Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALPPS (Experimental): ASSOCIATING LIVER PARTITION WITH PORTAL VEIN LIGATION FOR STAGED HEPATECTOMY (ALPPS)
  Associating Liver Partition and Portal Vein Ligation for Staged Hepatectomy (ALPPS) is performed according to local practice in the respective centers. Preconditions to participation are experience with major liver resections and documentation of having performed at least 5 ALPPS cases prior to participation due to the learning curve with this quite complex procedure.
  The amount of transsection (in-situ split/liver partition) in Step 1 is left to the participating center, no minimal % of transsection is specified.
  Interventions: Procedure: ALPPS
- TWO STAGE HEPATECTOMY (Active Comparator): TWO STAGE HEPATECTOMY (TSH)
  Two-Stage Hepatectomy is defined as:
  1. Partial resection + portal vein ligation (RES PVL)
  2. Partial resection + secondary portal vein embolization (RES PVE). Followed by (extended) hemihepatectomy after an interval to induce hypertrophy of the liver.
  Conventional Two- Stage Hepatectomies will be standard procedures of the centers participating in the study.
  Interventions: Procedure: TWO STAGE HEPATECTOMY

INTERVENTIONS:
Procedure: ALPPS — For detailed information please refer to description of experimental arm
  Other Names: Associating Liver Partition and Portal Vein Ligation for Staged Hepatectomy
  Arms: ALPPS
Procedure: TWO STAGE HEPATECTOMY — For detailed information please refer to description of active comparator arm
  Other Names: TSH
  Arms: TWO STAGE HEPATECTOMY

SUMMARY:
Surgical resection has offered the best option for prolonged survival in patients with colorectal liver metastases. Limiting factor for major liver resections is the size of the future liver remnant (FLR). In case of normal liver function, 30% of the total liver volume is considered to be sufficient to maintain adequate liver function after resection. In an attempt to further increase "resectability" criteria for patients with too small FLR surgical and interventional maneuvers such as portal vein embolization and portal vein ligation in two-stage hepatectomies have been implemented, but they need an interval of 4-8 weeks to achieve sufficient hypertrophy. In order to obtain adequate but rapid parenchymal hypertrophy a new surgical two-step technique, ALPPS, was introduced for oncological patients requiring extended hepatic resection with limited functional reserve. Both procedures can be performed with acceptable morbidity and mortality.

The investigators conclude that it is time to perform a randomized study comparing the two surgical approaches in regard to oncological outcome.

ELIGIBILITY:
Inclusion Criteria:

Patients fulfilling all of the following inclusion criteria may be enrolled in the study:

* Male or female patients above 18 years of age.
* Patients with multifocal CRLM with a FLR/TLV (Total Liver Volume)< 30% OR a FLR/BW (Bodyweight) ratio of < 0.5.
* Patients with colorectal primary tumor not yet resected may be included as long as the extrahepatic disease may be cured surgically (liver first strategy).
* Patients with lung metastases may be included in the study as long as the lung metastases are potentially curable by resection by judgment of a thoracic surgery consultant.
* Chemotherapy response according to RECIST: regression or stable disease.
* The indication for surgery should be discussed at a multidisciplinary tumor board attended by hepatobiliary surgeons, oncologists, hepatologists and radiologists.
* Written informed consent given by the patient after discussing the trial with the patient in a language he/she understands.
* For women of chlidbearing age: Not currently breastfeeding; usage of effective contraception if sexually active; not pregnant and agreement not to become pregnant during the 12 months thereafter. A negative pregnancy test before inclusion into the trial is required for women, who are not yet menopausal, had their last menses within less than 12 months or have not had uterus and or ovaries removed surgically or undergone tubal ligation.

Exclusion Criteria:

The presence of any one of the following exclusion criteria will lead to exclusion of the participant:

* Male or female patients under 18 years of age.
* Unilobar tumorload qualifying the subject for a standard hepatectomy.
* Patients with multifocal CRLM with a FLR/TLV > 30% OR a FLR/BW ratio of > 0.5.
* Patients with a baseline FLR of less than 15%.
* Patients with extrahepatic metastatic disease (except potentially resectable lung metastases).
* Patients not having received chemotherapy before study enrollment.
* If the liver biopsy prior to enrollment or the first liver biopsy in stage I shows fibrosis (Metavir stage ≥F3) or >30% macrosteatosis.
* Significant concomitant diseases making the patient unsuitable for major liver surgery by the judgment of the physicians involved.
* Known or suspected non-compliance (e.g. drug- and/or alcohol abuse).
* Enrollment into a clinical trial interfering with the endpoints.
* Intention to become pregnant during the course of the study.
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases.
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.
* Previous enrollment in the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
1 Year Disease-free Survival | 1 year after Randomization
  The primary objective will be disease-free survival at one year after randomization as determined by PET-CT (Positron emission tomography - Computer tomography), when not available by CT (Computer tomography) Thorax/Abdomen. This will be assessed by two independent radiologists who will be blinded to which arm the patient was enrolled in.
  Patients who died, are lost to follow up or are too sick to undergo imaging will be censored and counted as failures to reach the primary endpoint.
  Patients may need resection of their primary tumor after the study intervention (liver first strategy). They may develop recurrence within the study period, systemic or in the liver. In these patients ablation, reoperation and chemotherapy are used as customary clinical routine. Whether they achieved tumor free survival however depends only on the PET-CT or CT Thorax Abdomen at one year.

SECONDARY OUTCOMES:
Procedure-associated Mortality | Up to 1 year after Randomization
  All deaths will be recorded in the 12 month-period after randomization. Specifically, the number of patients, which suffer a fatal event due to the procedure during the postoperative period, will be calculated to assess the safety of the two interventions.
Procedure-associated Complications | Up to 1 year after Randomization
  Complications during the postoperative period will be recorded using the Clavien-Dindo Classification, also known as the Zurich Classification, which grades surgical Complications on a scale from 1 to 5 (death of patient).
  Dindo D, Demartines N, Clavien PA: Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13.
Percentage of patients in which complete curative two-staged surgery was possible. | Up to 1 year after Randomization
  The percentage of patients, in which a complete curative two-staged surgical procedure was possible, will be assessed.
  "Complete" is defined as successful completion of both surgical steps of the procedure, i.e.:
  * step 1: cleaning of tumorlesions in the future liver remnant (FLR) and portal vein ligation of the contralateral segments to induce hypertrophy of the FLR (with or without in situ split/transsection).
  * step 2: resection of the tumorbearing part of the liver, leaving a tumor-free FLR in situ.
  "Curative" is defined as achieving a tumorfree FLR after step 2 with no signs of extrahepatic tumor existance.
  (If patients have the primary tumor or potentially resectable lung metastases, which will be approached surgically in the future treatment of the patient in a curative intent, then the procedure does count as curative).
Complete (R0) vs. incomplete (R1/2) resection (oncological outcome) | 1 year after Randomization
  A consensus between pathologists and surgeons on the R-status of the resection, judging both stages separately and together. Through re-resection R0 may be achieved overall even if there was a R1 resection after stage 1.
Overall survival (oncological outcome) | Up to 10 years after Randomization
  From date of randomization until the date of death from any cause, assessed up to 10 years.
  Regular further follow up-visits after assessment of the primary endpoint at 1 year are planned 1.5, 2, 3, 5 and 10 years after Randomization.
Quality of Life (QoL) | Up to 1 year after Randomization
  Will be evaluated by the Visual Analogue Scale (VAS) for Quality of Life in Cancer.
  Visual Analogue Scale determines QoL on a scale of 1 (worst) to 10 (best).
  First Baseline Assessment before stage 1 procedure. Assessment after procedure step 1. Assessment before stage 2 procedure. Assessment after procedure step 2. Regular assessments during scheduled and unscheduled follow-up visits.
Radiographic liver volumetric changes | Up to 1 year after Randomization
  Volumetry 1 performed before stage 1 of procedure Volumetry 2 performed before stage 2 of procedure
  All volumetries are performed locally via magnet resonance Imaging or computertomography and reported into a respective volumetry Case Report Form (CRF).
Incidence of posthepatectomy liver failure | Up to 1 year after Randomization
  The incidence of posthepatectomy liver failure is assessed according to the definition and grading by the International Study Group of Liver Surgery (ISGLS), which separates 3 different grades of posthepatectomy liver failure (Grade A to C).
  Rahbari, N. N., et al. (2011). "Posthepatectomy liver failure: a definition and grading by the International Study Group of Liver Surgery (ISGLS)." Surgery 149(5): 713-724.
Incidence of posthepatectomy liver failure | Up to 1 year after Randomization
  The incidence of posthepatectomy liver failure is assessed according too the "50:50 Criteria".
  Balzan, S., et al. (2005). "The "50-50 criteria" on postoperative day 5: an accurate predictor of liver failure and death after hepatectomy." Ann Surg 242(6): 824-828, discussion 828-829.
Incidence of posthepatectomy renal failure | Up to 1 year after Randomization
  Measurement of the following parameter at screening visit, during the postoperative course of stage 1 & 2 (postoperative days 1,2,3,5,7) and at follow-up visits:
  * Creatinin [Unit: µmol/l]
  This parameter is used to calculate and assess the incidence of posthepatecomy renal failure according to the AKIN-criteria.
  Ricci, Z., et al. (2011). "Classification and staging of acute kidney injury: beyond the RIFLE and AKIN criteria." Nat Rev Nephrol 7(4): 201-208.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Alain Clavien, MD, PhD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No